CLINICAL TRIAL: NCT02895438
Title: Does Non Coeliac Gluten Sensitivity (NCGS) Exist in Children? A Double-Blind Randomized Placebo-Controlled Trial
Brief Title: Non Coeliac Gluten Sensitivity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1408204; 2015-A00060-49 (Other: ANSM)
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Diet, Gluten-Free; Gluten-Sensitive Enteropathy
Keywords: Gluten-Sensitive; Diet, Gluten-Free; Irritable Bowel Syndrome; non Coeliac Gluten sensitivity; children
MeSH Terms: conditions — Celiac Disease; Irritable Bowel Syndrome | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gluten (Experimental): One group had a introduction of gluten followed by a wash-out period, then a placebo introduction, whereas the other group had the placebo first, then the wash-out and the gluten introduction.
  Interventions: Dietary Supplement: gluten
- Placebo (Active Comparator): One group had a introduction of gluten followed by a wash-out period, then a placebo introduction, whereas the other group had the placebo first, then the wash-out and the gluten introduction.
  Interventions: Dietary Supplement: gluten

INTERVENTIONS:
Dietary Supplement: gluten

SUMMARY:
Irritable Bowel syndrome (IBS) is a very frequent condition in children. Its management is difficult, often resulting in a persistence of chronical abdominal pain.

In adults, many patients affected by IBS improve under a gluten-free diet, even in the absence of Celiac Disease (CD) or wheat allergy. This condition is called Non Coeliac Gluten Sensitivity (NCGS). However, it is still not clear how to diagnose and manage NCGS, and the pathophysiological mechanisms also remain elusive.

The aim of this study is to determine if NCGS exists in children with IBS and to identify the clinical, serological, and histological characteristics, which could distinguish patients with NCGS from conventional IBS and CD patients.

This is a prospective cohort study in a population of children affected by a moderate to severe IBS for more than 6 months. All children had a Gluten Free Diet (GFD) for 6 weeks. Then, children who improved under GFD were randomized in two groups for a double-blind placebo-controled trial. One group had a reintroduction of gluten followed by a wash-out period, then a placebo reintroduction, whereas the other group had the placebo first, then the wash-out and the gluten reintroduction.

ELIGIBILITY:
Inclusion Criteria:

* children with Irritable Bowel Syndrome (IBS)

Exclusion Criteria:

* children with Celiac Disease (CD)
* children with wheat allergy

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Severity of IBS | 12 weeks after randomisation
  assessed though the composite score of FRANCIS

SECONDARY OUTCOMES:
change in gastro-intestinal symptoms | 12 weeks after randomisation
  assessed by Visual Analog Scale
Change in quality of life | 12 weeks after randomisation
  assessed by PedsQL scale

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie DESTOMBE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No